CLINICAL TRIAL: NCT03688984
Title: A Randomized Controlled Trial of Cognitive-behavioural Therapy for Insomnia (CBT-I) for Adolescents With Mild Traumatic Brain Injury
Brief Title: Treatment of Insomnia for Adolescents With Mild Traumatic Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REB16-1166
Record Dates: First submitted 2018-09-13; First posted 2018-09-28 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Mild Traumatic Brain Injury; Post-Concussion Syndrome; Insomnia
MeSH Terms: conditions — Brain Concussion; Post-Concussion Syndrome; Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Assessors will be blind to randomization condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Behavioural Therapy for Insomnia (Experimental): Six sessions of in person Cognitive Behavioural Therapy for Insomnia (CBT-I)
  Interventions: Behavioral: Cognitive Behavioural Therapy for Insomnia
- Treatment As Usual (No Intervention): Participants will receive regular care in the Treatment As Usual (TAU) condition. Participants will be offered CBT-I at the completion of the trial.

INTERVENTIONS:
Behavioral: Cognitive Behavioural Therapy for Insomnia — Cognitive Behavioural Therapy for Insomnia (CBT-I) consists of six individual therapy sessions that last approximately one hour each. The sessions include psychoeducation about insomnia, goal setting, relaxation training, stimulus control, sleep consolidation and medication review. Additional components include cognitive therapy, sleep hygiene and mindfulness and relapse prevention.
  Arms: Cognitive Behavioural Therapy for Insomnia

SUMMARY:
A substantial number of children and adolescents sustain a mild traumatic brain injury (mTBI) each year. Although research supports that the vast majority of youth will recover quickly and return to normal functioning, some adolescents continue to report problems long after the injury. Disturbed sleep, notably trouble with sleep onset and sleep maintenance, is a frequently reported problem in those with slow recovery from a mTBI. Poor sleep is also associated with cognitive complaints, mood disturbance, and lower quality of life. Despite the identification of sleep disturbance as a problem associated with slow recovery, there are very few treatment options. Cognitive-behavioural therapy for insomnia (CBT-I) has shown promise in children and adolescents as an effective treatment for sleep disturbance, although it has yet to be applied to the adolescent mTBI population who also present with sleep problems. The objective of this study is to examine the treatment of sleep disturbance using cognitive-behavioural therapy for insomnia (CBT-I) in those adolescents who have a protracted recovery from their mTBI. This represents a novel treatment option for this patient population and is anticipated to improve outcomes and quality of life.

DETAILED DESCRIPTION:
Mild traumatic brain injuries (mTBIs) in youth are a major public health issue. The vast majority of adolescents who sustain a mTBI will recover within a few months. Epidemiological studies of youth with mTBI who present to the emergency department suggest that roughly 80-85% of school-aged children and adolescents will recover symptomatically by 3 months post-mTBI. These recovery rates suggest that only a small proportion of children with mTBI will show a protracted recovery. Unfortunately, these children require considerable health care resources, miss a large amount of academic time, and suffer declines in quality of life. There is a paucity of evidence-based treatment for the constellation of problems displayed by those with protracted recovery from mTBI, with most current practices focusing on amelioration of specific symptoms using pharmacological agents.

Following a mTBI, sleep disruption is a commonly reported symptom. Blinman and colleagues reported symptom characteristics in adolescents who were admitted to the hospital following a mTBI. When rating symptoms during the initial hospitalization, 55% reported having trouble falling asleep and 54% reported sleeping less than usual. When asked again 2-3 weeks follow-up, 38% reported having trouble falling asleep and 22% reported sleeping less than usual. Of the 22 symptoms being rated at the 2-3 week follow-up, sleep issues had some of the highest mean symptom severity ratings. Although sleep problems are often endorsed acutely after the injury, true sleep disturbance likely has a slightly delayed onset compared to physical symptoms (e.g., headaches, dizziness). Eisenberg and colleagues suggested that sleep problems resolved gradually over time, but evidence suggests that they can persist in a sub-sample of children with mTBI, particularly if the sleep difficulties arise early in recovery.

Cognitive behavioural therapy for insomnia (CBT-I) represents a promising therapeutic option for sleep disruption following mTBI in youth. Although sleep disturbance is a common post-concussive problem, few treatment options are available. CBT-I has been shown to successfully treat insomnia in multiple populations and has been recommended as a first-line treatment for insomnia, because it shows superior long-term symptom reduction in comparison to both benzodiazepine and non-benzodiazepine drugs. Furthermore, meta-analyses support the effectiveness of CBT-I, with medium to large effect sizes for CBT-I on measures of subjective sleep both at the end of treatment and on follow-up. CBT-I is theorized to work similarly in adult and adolescent populations. Evidence suggests that the gains made from CBT-I persist over time and include shorter latency to fall asleep, fewer times of waking after sleep onset, and better sleep efficiency, as well as secondary improvements in child-reported depression and anxiety.

Objective:

To determine if CBT-I (in-person) improves sleep in adolescents with protracted recovery following a mTBI.

Hypotheses:

Primarily, the investigators hypothesize that in-person CBT-I will result in significant improvements in subjectively reported insomnia for adolescents with mTBI, over and above treatment as usual.

Secondarily, the investigators hypothesize that in-person CBT-I will result in significant improvements in subjective sleep quality, dysfunctional beliefs about sleep, and sleep diary measures for adolescents with mTBI, over and above treatment as usual.

Method:

Participants: Participants 12-18 years of age who are slow to recover from a mTBI will be recruited from the ACH Brain Injury Clinic (Dr. Barlow, Lisette Lockyer, Lisa Bodell) and from the ACH Neuropsychology Service (Dr.Brooks).

Procedure: This will be a single-blind parallel-group RCT that will block sex (1:1 ratio). Those in the control group who have insomnia at week 13 can be entered into the treatment at that time. Participants will be randomized and will complete pre-treatment measures at week 1. The questionnaires are expected to take 30 minutes to complete (ISI, PSQI, DBAS, HBI, and PROMIS). Those randomized to the treatment arm (in-person CBT-I) will partake in a 6-week CBT-I program adapted for adolescents, with each session taking 1 hour. A breakdown of what each CBT-I session comprises is found in the study protocol. Sessions will be led by a postdoctoral fellow or graduate student overseen by Drs. Tomfohr-Madsen or Madsen (registered psychologists). Following treatment, participants will complete the same measures again. The same measures will be completed once more at one month post-treatment to measure maintenance of sleep improvement. The control group will participate in all assessment points, and may choose to partake in the CBT-I protocol after the final assessment if sleep problems persist.

This will be a randomized clinical trial - participants randomized to the treatment condition will partake in the CBT-I intervention. There is one treatment arm - in-person CBT-I. Participants randomized to the control condition may elect to partake in the CBT-I intervention following completion of all follow-up measures if their sleep problems persist.

Participants will complete pre-treatment measures at baseline (week 1). The questionnaires are expected to take 30 minutes for adolescents to complete (ISI, PSQI, DBAS-16, HBI, PROMIS depression and anxiety scales), plus 5 minutes daily for the sleep diary to be completed. Parents will provide demographic information (5-10 minutes). Those randomized to the treatment condition will partake in a 6-week CBT-I program (in-person) adapted for adolescents, with each session taking 1 hour. Corroboration of engagement in the treatment will be based on sleep diary entries. Sessions will be led by a postdoctoral fellow or graduate student overseen by Drs. Madsen and Tomfohr-Madsen (registered psychologists). Following the intervention, participants in both conditions will complete the same measures again at week 8 (assessors will be blinded to the study condition). The same measures will be completed one more time at one month post-treatment to measure maintenance of sleep improvement (assessors again blinded to study condition).

ELIGIBILITY:
Inclusion Criteria:

* 12-18 years of age
* diagnosed with a concussion by a nurse practitioner or physician at the ACH Complex Concussion Clinic (i.e., concussion was defined as an traumatic injury to the head, at least one reported symptom [e.g., dizziness, headache, nausea] at the time of the injury, and a Glasgow Coma Scale rating of ≥13/15 at 30 minutes after injury, or loss of consciousness <30 minutes, or post-traumatic amnesia <24 hours)
* being at least 2 months but no more than 12 months post-injury to ensure symptoms were no longer acute, yet current and persistent
* reporting elevated symptoms of insomnia measured by an Insomnia Severity Index score of ≥12
* ability to attend in-person treatment sessions.

Exclusion Criteria:

* moderate or severe TBI (i.e., Glasgow Coma scale rating of ≤12, loss of consciousness exceeding 30 minutes, and/or post-traumatic amnesia exceeding 24 hours)
* visual, hearing, motor, and/or language deficits that would hinder the completion of questionnaires or engagement in CBT-I.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2018-01-17 (Actual); Study Completion 2018-01-17 (Actual)

PRIMARY OUTCOMES:
Insomnia Severity Index (ISI) total score. | Baseline to post-treatment (7-weeks later)
  The ISI is a seven-item self-report questionnaire that assesses sleep onset latency, sleep efficiency, and functional impact from sleep issues. The sleep latency and efficiency items are rated on a 5-point Likert scale from 0 (none) to 4 (very severe). The remaining four items measure dissatisfaction, how noticeable sleep problems are to others, distress from sleep problems, and interference with daily functioning (all rated on 5-point Likert scales). Total scores on the ISI range from 0-28 with higher scores indicating more insomnia symptoms.

SECONDARY OUTCOMES:
Insomnia Severity Index (ISI) total score. | Baseline to follow-up (4-weeks later)
  The ISI is a seven-item self-report questionnaire that assesses sleep onset latency, sleep efficiency, and functional impact from sleep issues. The sleep latency and efficiency items are rated on a 5-point Likert scale from 0 (none) to 4 (very severe). The remaining four items measure dissatisfaction, how noticeable sleep problems are to others, distress from sleep problems, and interference with daily functioning (all rated on 5-point Likert scales). Total scores on the ISI range from 0-28 with higher scores indicating more insomnia symptoms.
Pittsburgh Sleep Quality Index (PSQI) Global Score | Baseline to post-treatment (7-weeks later) and a follow-up (4-weeks later)
  The PSQI is a widely used brief self-report measure of sleep quality aimed at examining the facets of sleep disturbance. It is composed of 19 items that measure sleep disruptions in the month prior to questionnaire completion. The PSQI contains seven subscales: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medications, and daytime dysfunction, which are combined into a total sleep quality score. The total PSQI raw score ranges from 0 to 21, with higher scores representing worse sleep disturbance; scores of greater than 5 indicate clinically significant sleep disruption.
Dysfunctional Beliefs about Sleep (DBAS-16) total score | Baseline to post-treatment (7-weeks later) and a follow-up (4-weeks later)
  The DBAS was developed to identify unhelpful beliefs about sleep, and is composed of 16 items organized on an 11-point Likert scale that ranges from 0 (strongly disagree) to 10 (strongly agree). All item scores are summed and averaged to calculate a total raw score where higher scores indicate more negative beliefs and attitudes towards sleep. Scores range from 0-10.
Total sleep time (TST) as assessed via 7-night sleep diary. | Baseline to post-treatment (7-weeks later) and a follow-up (4-weeks later)
  Participants completed an online sleep diary for the seven consecutive nights immediately following the completion of their questionnaire battery. Participants were asked to complete the sleep diary within an hour of waking up. The online sleep diary consisted of eight items assessing bedtime, duration of sleep initiation, night time waking, wake time, get-up time, nap time, and overall length and perceived quality of sleep.Across each of the 7-day assessment periods, average total sleep time (TST), wake after sleep onset (WASO), sleep onset latency (SOL) and sleep efficiency (SE) were calculated.
Wake after sleep onset (WASO) as assessed via 7-night sleep diary | Baseline to post-treatment (7-weeks later) and a follow-up (4-weeks later)
  Participants completed an online sleep diary for the seven consecutive nights immediately following the completion of their questionnaire battery. Participants were asked to complete the sleep diary within an hour of waking up. The online sleep diary consisted of eight items assessing bedtime, duration of sleep initiation, night time waking, wake time, get-up time, nap time, and overall length and perceived quality of sleep.Across each of the 7-day assessment periods, average total sleep time (TST), wake after sleep onset (WASO), sleep onset latency (SOL) and sleep efficiency (SE) were calculated.
Sleep onset latency (SOL) as assessed via 7-night sleep diary | Baseline to post-treatment (7-weeks later) and a follow-up (4-weeks later)
  Participants completed an online sleep diary for the seven consecutive nights immediately following the completion of their questionnaire battery. Participants were asked to complete the sleep diary within an hour of waking up. The online sleep diary consisted of eight items assessing bedtime, duration of sleep initiation, night time waking, wake time, get-up time, nap time, and overall length and perceived quality of sleep.Across each of the 7-day assessment periods, average total sleep time (TST), wake after sleep onset (WASO), sleep onset latency (SOL) and sleep efficiency (SE) were calculated.
Sleep efficiency (SE) as assessed via 7-night sleep diary | Baseline to post-treatment (7-weeks later) and a follow-up (4-weeks later)
  Participants completed an online sleep diary for the seven consecutive nights immediately following the completion of their questionnaire battery. Participants were asked to complete the sleep diary within an hour of waking up. The online sleep diary consisted of eight items assessing bedtime, duration of sleep initiation, night time waking, wake time, get-up time, nap time, and overall length and perceived quality of sleep.Across each of the 7-day assessment periods, average total sleep time (TST), wake after sleep onset (WASO), sleep onset latency (SOL) and sleep efficiency (SE) were calculated.
PROMIS® Depression Scale total score | Baseline to post-treatment (7-weeks later) and a follow-up (4-weeks later)
  The pediatric PROMIS® Depression questionnaire was developed by the NIH to evaluate symptoms of depression, such as feelings of hopelessness, helplessness, and worthlessness in pediatric populations. The self-report version of the PROMIS® Depression questionnaire was included in this study. This 8-item measure queries depression symptom presentation based on the past seven days, with each item rated on a 5-point Likert scale ranging from 1 (never) to 5 (almost always). All items were summed to calculate a total raw score where higher scores indicate more severe depressive mood. symptomology.
PROMIS® Anxiety Scale total score | Baseline to post-treatment (7-weeks later) and a follow-up (4-weeks later)
  The pediatric PROMIS® Anxiety questionnaire was developed by the National Institutes of Health (NIH) to evaluate symptoms of anxiety, such as feelings of fear, anxious misery, and hyperarousal in pediatric populations. The self-report version of the PROMIS® Anxiety questionnaire was included in this study. This 8-item measure queries anxiety symptom presentation based on the past seven days, with each item rated on a 5-point Likert scale ranging from 1 (never) to 5 (almost always). All item scores were summed to calculate a total raw score where higher scores indicate more severe anxiety symptomology.
Health and Behavior Inventory (HBI) total score | Baseline to post-treatment (7-weeks later) and a follow-up (4-weeks later)
  The Health and Behavior Inventory (HBI) was used to measure the presence and severity of post-concussive symptoms based on adolescent self-report. The HBI measures the frequency of common somatic and cognitive post-concussive complaints and does not include any sleep-related items. The HBI is a 20-item questionnaire where symptoms are rated on a 4-point Likert scale ranging from 1 (never) to 4 (often) based on frequency over the past week. All items were summed to calculate a total raw score where higher scores indicate more severe post-concussive symptoms. The HBI was developed as a measure for both child and parent-proxy reports of post-concussive symptoms in children.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Brooks, PhD, Principal Investigator — University of Calgary
Locations (1):
- Alberta Children's Hospital, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
Data wil be published by the primary study team.

REFERENCES:
- [Derived] Tomfohr-Madsen L, Madsen JW, Bonneville D, Virani S, Plourde V, Barlow KM, Yeates KO, Brooks BL. A Pilot Randomized Controlled Trial of Cognitive-Behavioral Therapy for Insomnia in Adolescents With Persistent Postconcussion Symptoms. J Head Trauma Rehabil. 2020 Mar/Apr;35(2):E103-E112. doi: 10.1097/HTR.0000000000000504. PMID 31246882

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-09-19): https://cdn.clinicaltrials.gov/large-docs/84/NCT03688984/Prot_SAP_ICF_000.pdf